CLINICAL TRIAL: NCT03297697
Title: A Multi-Institutional Prospective Cohort Study of Minimal Residual Disease in Peripheral T-cell Lymphoma
Brief Title: Minimal Residual Disease in Peripheral T-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Invivoscribe, Inc. (Industry); National Cancer Institute (NCI) (NIH); T-Cell Leukemia Lymphoma Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201706050; 5K12CA167540-07 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bone marrow, and tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Arm 1: Lymphotrack: -Patients will be treated with frontline chemotherapy per the treating physician's discretion. Collection of the pre-treatment tumor biopsy to identify the tumor-specific clonotype and peripheral blood samples at various time points for assessment of minimal residual disease using the LymphoTrack MRD assay. The results of these studies will be performed in batches and therefore will not be available to patients and clinicians to make clinical decisions.
  Interventions: Procedure: Tumor biopsy; Procedure: Peripheral blood draw; Procedure: Lymphotrack TCR clonality assay

INTERVENTIONS:
Procedure: Tumor biopsy — Biopsy specimen can be from bone marrow, blood, or lymph node. This specimen should have a high disease load
Procedure: Peripheral blood draw — -Baseline, C1D1, C1D8, C1D15, C2D1, C3D1, C4D1, C5D1, C6D1, end of treatment, 3 month follow-up (optional), 6 month follow-up, 9 month follow-up (optional), 12 month follow-up, 15 month follow-up (optional), 18 month follow-up, 21 month follow-up (optional), 24 month follow-up, and at relapse
Procedure: Lymphotrack TCR clonality assay — -Assay with high sensitivity that can be performed with peripheral blood

SUMMARY:
As T-cell receptor sequencing by LymphoTrack is an assay with high sensitivity that can be performed in peripheral blood, the investigators wish to evaluate the ability of this assay to predict which patients are at higher risk of relapse after initial therapy for peripheral T-cell lymphomas which is being given for curative intent. Additionally, as more is known about the ability of dynamic monitoring of cfDNA in B-cell lymphomas to predict relapse, the investigators wish to explore the use of this technology in T-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Histologically-confirmed peripheral T-cell lymphoma being treated with curative intent. Eligible histologies include, but are not limited to: peripheral T-cell lymphoma, not otherwise specified; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma, ALK negative; and anaplastic large cell lymphoma, ALK positive.
* Plan for treatment with frontline multi-agent anthracycline containing chemotherapy for curative intent (for example, CHOP, CHOEP, EPOCH). A frontline therapy program can include different sequential phases of treatment, including high-dose therapy and autologous stem cell transplantation.
* Availability of pre-treatment test specimen from bone marrow, blood, lymph node, or alternate site to identify tumor-specific clonotype, or willingness to undergo biopsy if sufficient tissue is not available at time of enrollment (e.g. 15 slides from fixed formalin-fixed paraffin embedded tumor tissue

  *Patients who have less than 15 slides of fixed formalin-fixed paraffin embedded tumor tissue may be considered for enrollment after discussion with the study principal investigator
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Receiving second line of therapy or greater.
* Diagnosis of primary cutaneous T-cell lymphoma, extranodal NK-cell lymphoma, acute T-cell lymphoma/leukemia, hepatosplenic T-cell lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with peripheral T cell lymphoma who are seen in clinics associated with the participating locations
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of LymphoTrack TCR clonality assay of evaluating minimal residual disease as measured by progression-free survival (PFS) at the completion of 2 years | 2 years

SECONDARY OUTCOMES:
Feasibility of LymphoTrack TCR clonality assay of evaluating minimal residual disease as measured by the ability of Lymphotrack to detect minimal residual disease in at least 60% of baseline samples | Baseline
Evaluate whether LymphoTrack TCR clonality assay can distinguish participants with peripheral T-cell lymphomas (PTCL) who are at risk of relapse | Through 2 years
Percentage of participants with a dominant tumor sequence identified from the pre-treatment test specimen | Baseline
Determine whether monitoring for the tumor-specific clone at minimal residual disease (MRD) level predicts response to treatment | Through 2 years
Rate of decline of the tumor specific sequence or sequences predict duration of response | Through 2 years
Characterize the lead time from MRD positivity to subsequent clinical relapse | Through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, M.D., Study Chair — Washington University School of Medicine
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu